CLINICAL TRIAL: NCT01712269
Title: Understanding the Role Obesity Plays in the Pathogenesis of Obstructive Sleep Apnea
Brief Title: Assessment of Sleep Apnea and Its Causes Before and After Weight Loss Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI and main Co-I (Dr Edwards) relocated locations
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Atul Malhotra, MD, Associate Professor, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BWH-2011P002188; 5K24HL093218 (NIH)
Record Dates: First submitted 2012-10-16; First posted 2012-10-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Weight-loss (bariatric) surgery (Experimental): All subjects enrolled will undergo bariatric surgery to assist weight-loss
  Interventions: Procedure: Weight-loss (bariatric) surgery

INTERVENTIONS:
Procedure: Weight-loss (bariatric) surgery — Subjects will undergo bariatric surgery which will assist weight loss

SUMMARY:
The central aim of this research project is to determine how the ever-growing problem of obesity in the western world contributes to the pathophysiology of obstructive sleep apnea (OSA). To complete this aim, the investigators will determine the impact of obesity on the mechanisms underlying OSA. This will be achieved by making physiological measurements of 4 physiological traits known to cause OSA as well as the patients sleep apnea severity, before and after weight-loss surgery (i.e. bariatric surgery).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by repetitive collapse or 'obstruction' of the pharyngeal airway during sleep. These obstructions result in repetitive hypopneas/apneas and cause intermittent hypoxia/hypercapnia, as well as surges in sympathetic activity. Such processes disturb normal sleep and impair neurocognitive function, often resulting in excessive daytime sleepiness and decreased quality of life. Furthermore, OSA is associated with cardiovascular morbidity and mortality, making OSA a major health concern. Obesity is categorically the major risk factor for OSA, with available data indicating a prevalence of 40% in obese men (BMI > 30kg/m2) and up to 90% in morbidly obese individuals (BMI > 40kg/m2). Given the prevalence of obesity has risen to epidemic proportions, with approximately 60% of adults considered overweight and 30% obese, it has become one of the world's leading health care concerns and research priorities. Importantly, as the prevalence of obesity continues to rise, so too does the number of individuals developing OSA. Surprisingly, despite the dominant role played by obesity in OSA pathogenesis, the precise mechanisms by which obesity leads to OSA are unclear

Current evidence suggests that OSA pathogenesis involves the interactions of at least four physiological traits comprising 1) the pharyngeal anatomy and its propensity towards collapse 2) the ability of the upper airway dilator muscles to activate and reopen the airway during sleep (i.e. neuromuscular compensation), 3) the arousal threshold from sleep (i.e. the propensity for hypopneas/apneas to lead to arousal and fragmented sleep) and 4) the stability of ventilatory feedback loop (i.e. loop gain). The potential mechanisms by which obesity may alter the four traits has to date not been carefully assessed. Specifically, obesity has been suggested to a) compromise the anatomy by decreasing the airway size and increasing its collapsibility, but it may also b) impair neuromuscular compensation by increasing the mechanical load placed on the upper airway muscles, c) increase the loop gain and destabilize breathing potentially via reductions in lung volume and increased chemosensitivity or d) increase the arousal threshold and thereby reduce the propensity to arouse from sleep which may offset some of the obesity-related deficits in the other traits. However, we do not know how obesity alters these four traits (in the same individual) and whether it involves predominantly one or several of the mechanistic pathways.

Therefore the aim of our study is to determine the impact of obesity on the mechanisms underlying OSA. This will be achieved by making physiological measurements before and after weight-loss surgery (i.e. bariatric surgery). Specifically we will assess:

1. The severity of OSA (apnea-hypopnea-index or AHI)
2. The physiological traits responsible for OSA:

i. Pharyngeal anatomy and its propensity towards collapse

ii. The ability of the upper airway dilator muscles to activate and reopen the airway during sleep (i.e. neuromuscular compensation).

iii. Arousal threshold from sleep (i.e. the propensity for hypopneas/apneas to lead to arousal and fragmented sleep).

iv. Stability of ventilatory feedback loop (i.e. loop gain).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 65 years
* BMI > 35kg/m2
* Scheduled for weight-loss surgery

Exclusion Criteria:

* Previous history of bariatric surgery
* Any serious medical condition (except controlled hypertension and diabetes)
* Any sleep disorder except OSA (RLS, insomnia, etc.)
* Use of medications known to affect sleep/arousal, breathing, or muscle physiology
* Allergy to lidocaine or Afrin
* History of current cigarette smoking or previous smoking history >10 pack years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-10; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Model prediction of absence/presence of OSA | Subjects will be assessed at baseline (pre-surgery)
  Our published method estimates 4 important physiological traits causing OSA: 1) pharyngeal anatomy, 2) loop gain, 3) the ability of the upper airway to dilate/stiffen in response to increases in ventilatory drive, and 4) arousal threshold. These variables are measured using a single maneuver in which CPAP is dropped from an optimum to various suboptimum pressures during sleep. Each individual's set of traits is then entered into a physiological model of OSA that graphically illustrates the relative importance of each trait in that individual and predicts OSA presence/absence.
Model prediction of absence/presence of OSA | Subjects will be assessed between 9-12 months post surgery
  Our published method estimates 4 important physiological traits causing OSA: 1) pharyngeal anatomy, 2) loop gain, 3) the ability of the upper airway to dilate/stiffen in response to increases in ventilatory drive, and 4) arousal threshold. These variables are measured using a single maneuver in which CPAP is dropped from an optimum to various suboptimum pressures during sleep. Each individual's set of traits is then entered into a physiological model of OSA that graphically illustrates the relative importance of each trait in that individual and predicts OSA presence/absence.

SECONDARY OUTCOMES:
Apnea-Hypopnea Index | Subjects will be assessed at baseline (pre-surgery)
  The Apnea-Hypopnea Index (AHI) is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow)
Apnea-Hypopnea Index | Subjects will be assessed between 9-12 months post surgery
  The Apnea-Hypopnea Index (AHI) is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Malhotra, MD, Principal Investigator — Brigham & Womens Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No